CLINICAL TRIAL: NCT02106858
Title: Stivarga® Regulatory Post-Marketing Surveillance Study in Korea
Brief Title: Stivarga Regulatory Post-Marketing Surveillance Study in Korea
Acronym: StivargaPMS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16778; SV1314KR (Other: Company Internal)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Neoplasms
Keywords: Stivarga / Regorafenib / Metastatic Colorectal Cancer / Metastatic or unresectable locally advanced GIST (Gastrointestinal stromal tumors)
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients treated by Physician with Stivarga under approved local prescriptions
  Interventions: Drug: Regorafenib (Stivarga,BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga,BAY73-4506) — Patients treated by Physician with Stivarga under approved local prescriptions

SUMMARY:
To investigate and collect post-marketing data on the safety of Stivarga in real world practice in its registered indication(s) as required by Health Authority.

ELIGIBILITY:
* Inclusion Criteria:
* Signed and dated informed consent
* Patients diagnosed with histologically confirmed metastatic colorectal cancer and/or metastatic or unresectable locally advanced gastrointestinal stromal tumors and/or HCC who have been previously treated with sorafenib by physician
* Patients who are prescribed with Stivarga tablet 40mg(Regorafenib) for the first time
* Exclusion Criteria:
* Patients participating in an investigational program with interventions outside of routine clinical practice
* All contra-indications according to the local marketing authorization have to be considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with metastatic colorectal cancer or metastatic or unresectable locally advanced GIST(Gastrointestinal stromal tumors) by physician.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with serious adverse events | Up to 30 days after terminating treatment
  Every 2 months (monthly safety assessment within first two cycles)
Percentage of patients with adverse drug reactions (ADRs) | Up to 30 days after terminating treatment
  Every 2 months (monthly safety assessment within first two cycles)

SECONDARY OUTCOMES:
Overall response | Up to 6 years
Progression free survival (PFS) | Up to 6 years
Overall survival (OS) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, South Korea